CLINICAL TRIAL: NCT05642052
Title: Feasibility Study of a Community Pilot Project for the Prevention of Alzheimer's Disease: the KetoHome Study.
Acronym: KetoHome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Nestlé Health Science (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-4327
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Alzheimer Disease; Glucose Metabolism
Keywords: Nutritional intervention; Glucose monitoring; Reduced carb diet; Energy metabolism; Ketones
MeSH Terms: conditions — Alzheimer Disease; Ketosis | interventions — Diet

STUDY DESIGN:
Intervention Model Description: All participants will go through 10 days of control diet and 10 days of reduced carb diet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 days control diet (Sham Comparator): Participants stay on their regular diet while glucose is continuously monitored, heart rate and number of steps is measured for 10 days.
  Interventions: Dietary Supplement: Regular diet
- 10 days low carb diet (Active Comparator): Participants will eat a low carb diet while glucose is continuously monitored, heart rate and number of steps is measured for 10 days.
  Interventions: Dietary Supplement: low carb diet

INTERVENTIONS:
Dietary Supplement: low carb diet — low carb meals will be 50% less carbs than the regular meals
  Other Names: reduced carb menu
  Arms: 10 days low carb diet
Dietary Supplement: Regular diet — Regular diet
  Other Names: Control
  Arms: 10 days control diet

SUMMARY:
The purpose of this study is to assess whether it is possible to carry out a research project with a nutritional intervention in senior's residence. Life in a small community is very different and above all unique, which could be an asset in a research setting.

DETAILED DESCRIPTION:
To ensure its functioning, the brain needs a lot of energy. However, during aging, it has difficulty properly using its main fuel, sugar. The brain then becomes "starved". This energy deficit is part of the vicious circle leading to memory problems. The brain, like a hybrid car, can run on two fuels, sugar and ketones. Providing alternative fuel to the brain, in the form of ketones, and thus offsetting the energy it needs, could improve its functioning and help prevent or improve memory problems.

There are several ways to increase ketones in our body such as certain dietary oils, natural health products, physical activity or certain diets. Reducing the amount of sugar in our diet is also a strategy that can increase ketones. A low-sugar diet is already widely used in the prevention of several important diseases, including type 2 diabetes and even Alzheimer's disease.

This study will assess the feasibility of a community intervention project in a seniors' residence with the eventual overall objective of slowing the progression or onset of AD and related health indicators, through a dietary modification.

This feasibility study will last 6 months. The basic characteristics of interested participants will be collected. The global spheres of evaluation are the following: metabolic profile, cognition, quality of life and nutritional status. Glucose measurements will be taken continuously via a sensor over two weeks during the project.

ELIGIBILITY:
Inclusion Criteria:

* Older men or women resident of Grace Village and resident of Vü;
* Understand, read and write French or English;
* Possess sufficient visual and auditory acuity to pass the cognitive tests.

Exclusion Criteria:

* The minimum possible criteria ensuring the safety of voluntary participants. The family doctor will need to confirm eligibility.
* Body mass index < 22
* Malnutrition.
* High risk of hypoglycaemia
* Moderate to severe digestive diseases that can be aggravated by dietary changes
* Severe dysphagia
* Supplementation with MCT oil, ketone salts, ketone ester, adherence to the ketogenic diet, intermittent fasting, or other diet or supplements that may significantly increase ketones;
* Participation in other intervention research projects on nutrition or aimed at metabolic change simultaneously.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Blood glucose concentrations | over 10 days
  in mmol/L

SECONDARY OUTCOMES:
Heart rate | 8 hours a day during 10 days
  beats per minutes
Number of steps | 8 hours a day during 10 days

OTHER OUTCOMES:
Menu appreciation level | After le 10 days of low carb diet
  To measure feasibility of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Rearsh Centre on Aging, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No